CLINICAL TRIAL: NCT03269903
Title: TTS Esophageal HILZO Covered Self-expandable Metal Stent for Palliation of Malignant Dysphagia: A Safety and Feasibility Study
Brief Title: TTS Esophageal HILZO Stent: A Safety and Feasibility Study
Acronym: HILZO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Kebomed B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL.59951.091.16
Record Dates: First submitted 2017-05-29; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-05

CONDITIONS: Esophagus Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: Multicenter non-randomized prospective clinical study in 30 patients with malignant dysphagia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental): Patients with malignant dysphagia treated with the HILZO stent
  Interventions: Device: HILZO esophageal stent

INTERVENTIONS:
Device: HILZO esophageal stent — A fully covered esophageal self-expandable metal stent for malignant dysphagia

SUMMARY:
A multicenter non-randomized prospective clinical study assessing the safety and feasibility of the esophageal through-the-scope HILZO Covered self-expandable metal stent placement for palliation of malignant dysphagia

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the safety and efficacy of placement of the esophageal HILZO Covered stent with the TTS method in patients with non-operable malignant obstruction of the esophagus or esophagogastric junction, extrinsic malignant compression, or recurrent malignant dysphagia after esophagectomy.

Other (secondary) objects are to assess the effect of the stent on the presence of hyperplastic reaction after implantation, the functional complications and survival.

ELIGIBILITY:
Inclusion Criteria:

* Non-operable malignant obstruction of the esophagus or esophagogastric junction, extrinsic malignant compression, or recurrent malignant dysphagia after esophagectomy. A tumor is considered inoperable if the patient has local tumor infiltration in the surrounding organs, distant metastases or a poor general health due to serious concomitant disease. OR
* Recurrent dysphagia after prior radiation with curative or palliative intent for esophageal or gastric cardia cancer.
* Requiring treatment for dysphagia (dysphagia score of ≥ 2, according to Ogilvie2)
* Written informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Inappropriate cultural level and understanding of the study.
* Simultaneous participation in another clinical study
* Life expectancy of less than 12 months
* Stenosis after laryngectomy, or if the distance between the upper edge of the stent is less than 2 cm from the upper esophageal sphincter
* Tumor length of more than 12cm
* Previous stent placement for the same condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment associated adverse events during follow-up (safety) | 1 year
  Short term (within 7 days after treatment) and long term (after 7 days) major complications and minor complications. Major complications are defined as life threatening and severe complications such as perforation, haemorrhage, fistula formation and severe pain. Minor complications are defined as non-life threatening or moderately severe pain and gastroesophageal reflux.
Through-the-scope stent placement (feasibility): (1) ease of deployment at intended esophageal location | 1 day
  Technical success is defined as ease of through-the-scope deployment and placement of the stent at the required esophageal location.
Through-the-scope stent placement (feasibility): incidence of device related adverse device events at moment of stent placement | 1 day
  Device related adverse events are defined as all adverse events that take place during the through-the-scope stent placement. The incidence of the device related adverse events will be recorded.

SECONDARY OUTCOMES:
Dysphagia, measured with the Ogilvie Dysphagia score (functional outcome) | 6 months
  Ogilvie dysphagia score measured at: baseline, 2 weeks and every 4 weeks until death/stent removal, or until a maximum of 6 months follow-up.
Retrosternal pain related to esophageal stent, measured with the Visual Analog Scale (functional outcome) | 6 months
  Retrosternal pain related to esophageal stent, measured with the Visual Analog Scale. Measurements will take place at 2 weeks and every 4 weeks until death/stent removal, or until a maximum of 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Peter Siersema, professor, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vermeulen BD, Reijm AN, van der Bogt RD, van Hooft JE, Spaander MCW, Siersema PD. Through-the-scope placement of a fully covered metal stent for palliation of malignant dysphagia: a prospective cohort study (with video). Gastrointest Endosc. 2019 Dec;90(6):972-979. doi: 10.1016/j.gie.2019.06.030. Epub 2019 Jun 29. PMID 31265819